CLINICAL TRIAL: NCT02669875
Title: Serelaxin To Lower Portal Pressure in Patients With Cirrhosis and Portal Hypertension
Brief Title: Serelaxin To Lower Portal Pressure
Acronym: STOPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Novartis Pharmaceuticals (Industry); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STOPP
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Liver Cirrhosis; Hypertension, Portal
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — serelaxin protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serelaxin (Active Comparator): IV infusion of serelaxin (RLX030) for 2 hours
  Interventions: Drug: Serelaxin
- Placebo (Placebo Comparator): IV infusion of placebo (20mM sodium acetate pH5) matched to serelaxin for 2 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Serelaxin — Serelaxin solution diluted in 5% glucose volume/volume (v/v) solution
  Other Names: RLX030; Recombinant human relaxin-2
  Arms: Serelaxin
Drug: Placebo — Placebo solution (20mM sodium acetate pH5) diluted in 5% v/v glucose solution
  Arms: Placebo

SUMMARY:
Portal hypertension (an increase in blood pressure in the portal vein that carries the blood from the intestine and spleen to the liver) underlies most of the serious complications of liver cirrhosis. This randomised placebo controlled study in people with liver cirrhosis evaluates the acute effects serelaxin (RLX030) infusion on portal hypertension and liver blood flow.

DETAILED DESCRIPTION:
This study will investigate the effects of the investigational drug serelaxin (a recombinant form of the peptide human relaxin-2) on portal hypertension in patients with liver cirrhosis. The investigators will measure portal pressure by hepatic venous pressure gradient (HVPG) and hepatic blood flow by indocyanine green (ICG) clearance to evaluate the potential benefits of the drug. In a recently completed small exploratory open-label phase 2 study (EudraCT no. 201200023626, NCT01640964), Part B demonstrated that serelaxin can lower portal pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult subjects over 18 years of age
2. Able to provide written informed consent and able to understand and willing to comply with the requirements of the study
3. Clinical imaging-diagnosed or biopsy-proven liver cirrhosis of any aetiology
4. Evidence of portal hypertension either on imaging or previous endoscopy
5. Patients with large/grade 3 varices as identified by endoscopy within 6 months of screening must be in an endoscopic band ligation programme at the time of study entry
6. Suspected hepatic venous pressure gradient (HVPG) ≥10 mmHg at baseline

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Women of child-bearing potential not using highly effective methods of contraception
3. Severe liver failure defined by one of the following: Prothrombin activity <40%, Bilirubin >5 mg/dL (85umol/L), hepatic encephalopathy > grade I
4. A history of variceal bleed within 1 month prior to visit 1
5. Presence of any non-controlled and clinically significant disease that could affect the study outcome or that would place the patient at undue risk
6. Hepatocellular carcinoma or history of malignancy of any organ system (other than localized basal cell carcinoma of the skin) treated or untreated
7. Portal vein thrombosis
8. Previous surgical shunt or TIPSS
9. Current use of beta-blockers or nitrates, any other drug therapy known to have an influence on portal pressure (diuretics permitted provided patients have been on a stable dose for at least 30 days)
10. History of drug or alcohol abuse within 1 month of enrolment
11. Sitting Systolic Blood Pressure <110 mmHg at screening visit or within 10 minutes prior to starting study drug infusion
12. Use of other investigational drugs within 5 half-lives of enrolment, or within 30 days/until the expected pharmacodynamic effect has returned to baseline, whichever is longer
13. Significant arrhythmias, which include any of the following: sustained ventricular tachycardia, bradycardia with sustained ventricular rate < 45 beats per minute or atrial fibrillation/flutter with sustained ventricular response of > 90 beats per minute at rest, or Long QT syndrome or corrected QT interval (QTc) > 450 msec (QT correction will be performed using the Fridericia correction method: QTcF = QT/RR0.33) for males and > 460 msec for females at screening visit
14. Documented hypersensitivity to intravenous contrast agents and/or iodine
15. Severe renal impairment (eGFR<30mL/min /1.73m2)
16. Significant left ventricular outflow tract obstructions (e.g., severe valvular aortic stenosis, obstructive cardiomyopathy), severe mitral stenosis, restrictive amyloid myocardiopathy, acute myocarditis
17. Severe aortic insufficiency or severe mitral regurgitation for which surgical or percutaneous intervention is indicated
18. Major neurologic event including cerebrovascular events, within 30 days prior to screening
19. Clinical evidence of acute coronary syndrome currently or within 30 days prior to enrolment
20. History of hypersensitivity to study drug serelaxin or study drug ingredients
21. Inability to follow instructions or comply with follow-up procedures.
22. Permanent pacemaker, cardiac resynchronisation device or implantable cardioverter-defibrillator in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fasting hepatic venous pressure gradient (HVPG) | Baseline, after 2 hours

SECONDARY OUTCOMES:
Change from baseline in fasting hepatic venous pressure gradient (HVPG) | Baseline, after 1 hour
Change from baseline in fasting hepatic blood flow | Baseline, after 2 hours
  Measured from the concentration of indocyanine green (ICG) in the hepatic venous blood vs peripheral venous blood using the Fick Principle
Change from baseline in inferior vena cava pressure | Baseline, after 2 hours
Change from baseline in cardiac index | Baseline, after 2 hours
Change from baseline in systemic vascular resistance index | Baseline, after 2 hours
Number of participants with adverse events | 4 weeks
  Adverse events (AE) reporting will be summarized based on number of patients reported with abnormal laboratory values, clinically significant AE, serious adverse events or death
Change from baseline in blood biomarker measurements | Baseline, after 2 hours
Change from baseline in aortic pulse wave velocity | Baseline, after 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Unit, Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fallowfield JA, Hayden AL, Snowdon VK, Aucott RL, Stutchfield BM, Mole DJ, Pellicoro A, Gordon-Walker TT, Henke A, Schrader J, Trivedi PJ, Princivalle M, Forbes SJ, Collins JE, Iredale JP. Relaxin modulates human and rat hepatic myofibroblast function and ameliorates portal hypertension in vivo. Hepatology. 2014 Apr;59(4):1492-504. doi: 10.1002/hep.26627. Epub 2014 Mar 3. PMID 23873655
- [Background] Kobalava Z, Villevalde S, Kotovskaya Y, Hinrichsen H, Petersen-Sylla M, Zaehringer A, Pang Y, Rajman I, Canadi J, Dahlke M, Lloyd P, Halabi A. Pharmacokinetics of serelaxin in patients with hepatic impairment: a single-dose, open-label, parallel group study. Br J Clin Pharmacol. 2015 Jun;79(6):937-45. doi: 10.1111/bcp.12572. PMID 25511105
- [Derived] Gifford FJ, Dunne PDJ, Weir G, Ireland H, Graham C, Tuck S, Hayes PC, Fallowfield JA. A phase 2 randomised controlled trial of serelaxin to lower portal pressure in cirrhosis (STOPP). Trials. 2020 Mar 12;21(1):260. doi: 10.1186/s13063-020-4203-9. PMID 32164767